CLINICAL TRIAL: NCT07013942
Title: Additional Effects of Dry Needling With PNF on Spasticity and Functional Performance in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/80
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Spasticity; Dry Needling; Functional Performance
Keywords: Spasticity; stroke; dry needling; functional performance; EMG; Fugl meyer; Modified Ashworth scale
MeSH Terms: conditions — Muscle Spasticity; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling group (Experimental): This group will receive dry needling twice a week along with gait training, functional training. the aim of this is to reduce spasticity with the help of dry needling with will aid in the improvement by increasing the functionality of the affected limb. Dry needling will be performed twice a week along with the exercise program
  Interventions: Procedure: Dry Needling Group
- Sham needling group (Experimental): This group focuses on elimination or accounting the placebo effect that may surround the concept of dry needling, this group doesn't really receive dry needling however the illusion is created in addition to the functional training gait training that the patient is receiving, sham needling will be done twice a week along with the exercise program
  Interventions: Procedure: Sham Needling Group

INTERVENTIONS:
Procedure: Dry Needling Group — Group A, which will be considered the interventional group. This group will be receiving the dry needling along with the PNF techniques for spasticity and functional performance.
  Arms: Dry needling group
Procedure: Sham Needling Group — Group B, which will be considered the control group. This group will be receiving sham needling in addition to the PNF techniques for spasticity and the functional performance
  Arms: Sham needling group

SUMMARY:
Stroke is a prevalent cause of long-term disability, with a rising global incidence. Stroke patients commonly experience impaired balance and trunk control, which limits their daily activities and quality of life. Spasticity is the result of upper motor neuron lesion in which the reflex arc is spared, however there is a lesion to the descending pathways of the spinal cord, which leads to the hyper excitability of the alpha motor neurons. Spasticity is a form of velocity dependent hypertonia. When dry needle is applied it induces relaxation in the muscle by increasing the distance between the z lines in the sarcomere and reduces the overlapping of contractile proteins, which ultimately leads to relaxation in the muscle. Dry needling also reduces the firing of the afferent pathways from the local muscle to the spinal cord reducing the excitability of the alpha motor neurons this leads to reduce spasticity. A randomized control trial will be conducted in multidisciplinary lab of FUCP, department of physical medicine and rehabilitation of Fauji Foundation Hospital on the sample of 30 participants. The subjects will be randomized into two groups by sealed opaque envelope method. A treatment over the course of 6 weeks will be provided. Interventional group will be receiving dry needling in addition to Proprioceptive Neuromuscular Facilitation while the control group will receive sham needling in addition to Proprioceptive Neuromuscular Facilitation. Exercise training would be done for a total of 6 weeks, with needling twice a week, the session will last 30- 50 minutes. Using SPSS version 21 would do analysis. Ethical approval will be obtained from ERC of FUSH. Informed written consent will be obtained from all participants.

DETAILED DESCRIPTION:
* To determine the effects of balance training with and without gaze stability exercises on mobility in older adults with mild cognitive impairment. To determine the additional effects of dry needling with Proprioceptive neuromuscular facilitation in comparison to sham needling with proprioceptive neuromuscular facilitation on spasticity in stroke.
* To determine the effects of dry needling with Proprioceptive neuromuscular facilitation techniques in comparison to sham needling with proprioceptive neuromuscular facilitation on functional performance in stroke

ELIGIBILITY:
Inclusion Criteria:

* 18 years to 65 years of age.
* Males and females
* Post stroke spasticity
* Ischemic stroke

Exclusion Criteria:

* Non-compliant Diabetic patients
* Active Hypertensive patients
* Immuno compromised patients
* Patients with underlying infections
* Patients with autoimmune diseases
* Patients that have any contagious conditions

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Spasticity | 6 weeks
  EMG will be used to highlight spasticity. The increased values of the ratio indicates increased hyper excitability of neurons hence indicating higher spasticity and hypertonia. Reduction of this ratio indicates relaxation of the muscles and decreased hyper excitability of the afferent pathway
Functional Performance | 6 weeks
  Functional performance will be checked using Fugl meyer. The overall score is 226. Higher scores indicate better functional performances. And lower scores indicate functional limitations

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan